CLINICAL TRIAL: NCT04638920
Title: Molecular Breath Print of COPD Patients With Exacerbations Despite Triple Inhalational Therapy (TripleEX)
Brief Title: Molecular Breath Print of COPD Patients With Exacerbations Despite Triple Inhalational Therapy
Acronym: TripleEX
Status: Completed | Type: Observational
Sponsor: Malcolm Kohler (Other)
Collaborators: Deep Breath Intelligence (DBI) (Unknown)
Responsible Party: Sponsor-Investigator, Malcolm Kohler, Prof. Dr. med., University of Zurich
Organization: University of Zurich (Other)
Other Study IDs: BASEC-Nr. 2020-01954
Record Dates: First submitted 2020-11-16; First posted 2020-11-20 (Actual); Results first posted 2025-04-02 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: COPD Exacerbation
Keywords: Exhaled breath analysis; Mass spectrometry

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Exacerbators: Patients with acute COPD exacerbation under triple inhalation therapy
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Determination of specific molecular breath patterns by secondary electrospray ionization mass spectrometry (SESIHRMS) during and 8 weeks after a COPD exacerbation. Furthermore, breath patterns will be assessed for correlation and association with clinical outcomes and treatment.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* age >= 18 years
* staged according to GOLD recommendations
* GOLD stage 2-4, GOLD ABE classification
* hospitalization due to COPD exacerbation
* subjects adherent to triple inhalational therapy (beta-2-sympathomimetics, anticholinergics, steroids)
* suitable for follow-up assessment
* <48 hours after initiation of antibiotic therapy or systemic steroid therapy

Exclusion Criteria:

* physical or intellectual impairment precluding informed consent or protocol adherence
* known pregnancy
* congenital defects with direct impact on central metabolism e.g. amino acid metabolism defect
* uncontrolled diabetes (e.g. HbA1c >11% or Glc >20mmol/l)
* acute or chronic pulmonary disease other than COPD
* renal failure or renal replacement therapy (GFR < 15 mL/min)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with COPD (staged according to GOLD recommendations, aged ≥18 years) on adherent triple inhalational therapy, hospitalized due to COPD exacerbation
Sampling Method: Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2020-11-16 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Zurich, Zurich, Canton of Zurich, Switzerland

REFERENCES:
- [Derived] Sievi NA, Schmidt F, Fricke K, Baur DM, Basler S, Herth J, Kohler M. Acute COPD exacerbation despite triple inhaled therapy: a molecular insight - TripleEx study. Respir Res. 2025 Sep 26;26(1):273. doi: 10.1186/s12931-025-03352-0. PMID 41013424

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited at the University Hospital Zurich between November 2020 and April 2024. Study duration was extended due to lack of sufficient patients until July 2023.
Groups:
- Exacerbators: Patients with acute exacerbation of COPD under triple exhalation therapy
Period: Overall Study
Arm/Group | Exacerbators
Started | 35
Completed | 30
Not Completed | 5
Not completed — Withdrawal by Subject | 5

BASELINE CHARACTERISTICS:
Population: Data of 28 participants were included in the final analysis as five patients withdrew their participation and the main outcome (breath analysis) of two participants was not analyzable.
Arm/Group | Exacerbators
Number analyzed (Participants) | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 65 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 27
  Unknown or Not Reported | 0
GOLD ABE classification [Count of Participants; unit: Participants] — The classification incorporates patients' symptomatic assessemetn and risk of exacerbation. Class A shows less symptoms and 0 to 1 moderate exacerbation in the previous year. Class B shows high symptoms and 0 to 1 moderate exacerbation in the previous year. Class E shows high symptoms and ≥ 2 moderate exacerbations or ≥ 1 leading to hospitalization.
  Participants
    Class A | 1
    Class B | 4
    Class E | 23
Exacerbation history [Mean (Standard Deviation); unit: events] — acute COPD exacerbation history in the previous year
  events
    Number of acute COPD exacerbations | 1.3 (0.9)
    Number of severe acute COPD exacerbations | 1.0 (0.7)
Treatment during acute COPD exacerbation [Count of Participants; unit: Participants]
  Antibiotics only | 4
  Systemic corticosteroids only | 5
  Antibiotics and systemic corticosteroids | 19

OUTCOME MEASURES:

1. Primary Outcome: Change in Exhaled Breath Metabolites
Description: Number of exhaled breath features/metabolites that show a change in intensity (unit of features: mass over charge ratio) during vs after COPD exacerbation. Exhaled breath features are measured via mass spectrometer. Change is calculated as feature intensity during COPD exacerbation minus feature intensity after COPD exacerbation (8 weeks after) for each detected exhaled breath feature.
Time Frame: twice during 8 weeks
Population: Exhaled breath data of two participants were not analazable due to technical problems.
Measure: Number; unit: breath metabolites
Arm/Group | Exacerbators
Number analyzed (Participants) | 28
breath metabolites | 3298

2. Secondary Outcome: Symptoms
Description: Correlation of breath metabolites with symptoms (mMRC and CAT) both measured twice during and after COPD exacerbation
Time Frame: twice during 8 weeks
Reporting Status: Not Posted

3. Secondary Outcome: Inflammation
Description: Correlation of breath metabolites with CRP, eosinophils, and exhaled NO, all measured twice during and after COPD exacerbation
Time Frame: twice during 8 weeks
Reporting Status: Not Posted

4. Secondary Outcome: Causative Agents
Description: Correlation of breath metabolites with sputum microbiology and viral swabs, both measured twice during and after COPD exacerbation
Time Frame: twice during 8 weeks
Reporting Status: Not Posted

5. Secondary Outcome: Treatment
Description: Correlation of breath metabolites with inhalational drugs, steroids, and antibiotics, both measured during COPD exacerbation
Time Frame: measured once during COPD exacerbation
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Serious events were collected during study period between time of inclusion (acute COPD exacerbation) and follow-up visit at stable state approximately 8 weeks after inclusion.
Description: Serious event were defined as follows:
  Any unfavorable event where it cannot be excluded that the event is attributable to the sampling of biological material or the collection of health-related personal data, and which:
  1. requires inpatient treatment not envisaged in the project plan or extends a current hospital stay;
  2. results in permanent or significant incapacity or disability; or
  3. is life-threatening or results in death.
Arm/Group | Exacerbators
All-Cause Mortality (participants affected / at risk) | 0/35
Serious Adverse Events (participants affected / at risk) | 0/35
Other Adverse Events (participants affected / at risk) | 0/35

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-09-02): https://cdn.clinicaltrials.gov/large-docs/20/NCT04638920/Prot_SAP_000.pdf